CLINICAL TRIAL: NCT06241950
Title: An Open-Label, Systemic Gene Delivery Study to Evaluate the Safety, Tolerability and Expression of SRP-9001 in Association With Imlifidase in Subjects With Duchenne Muscular Dystrophy With Pre-existing Antibodies to rAAVrh74
Brief Title: A Gene Transfer Therapy Study to Evaluate the Safety and Efficacy of Delandistrogene Moxeparvovec (SRP-9001) Following Imlifidase Infusion in Participants With Duchenne Muscular Dystrophy (DMD) Determined to Have Pre-existing Antibodies to Recombinant Adeno-Associated Virus Serotype (rAAVrh74)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is being terminated due to a business decision.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9001-104; 2022-003407-15 (EudraCT Number)
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Gene-Delivery; DMD; Ambulatory; Pediatric; Duchenne; Pre-existing antibodies; rAAVrh74 Antibody; Seropositive; Seropositivity; Titer
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Delandistrogene Moxeparvovec after Imlifidase Infusion (Experimental): Participants may receive 1 or 2 doses of imlifidase, depending on rAAVrh74 antibody titer results. Then, based on their rAAVrh74 antibody titer, eligible participants may receive 1 dose of delandistrogene moxeparvovec infusion.
  Interventions: Genetic: delandistrogene moxeparvovec; Biological: imlifidase

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS
Biological: imlifidase — IV infusion of Imliﬁdase
  Other Names: Idefirix

SUMMARY:
This is a gene transfer therapy study evaluating the safety of delandistrogene moxeparvovec and delandistrogene moxeparvovec dystrophin expression in association with imlifidase, in participants with DMD with pre-existing antibodies to rAAVrh74 over a period of 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory per protocol specified criteria.
* Has a definitive diagnosis of DMD prior to Screening based on documentation of clinical findings and confirmatory genetic testing.
* Ability to cooperate with motor assessment testing.
* Has elevated rAAVrh74 antibody titers per protocol-specified requirements.
* A pathogenic frameshift mutation, nonsense mutation or premature stop codon or pathogenic variant in the DMD gene that is expected to lead to absence of dystrophin protein.
* Stable daily dose of oral corticosteroids for at least 12 weeks prior to Screening, and the dose is expected to remain constant throughout the study (except for modifications to accommodate changes in weight).

Exclusion Criteria:

* Previous treatment with imlifidase.
* Presence of any other clinically significant illness, including cardiac, pulmonary, hepatic, renal, hematologic, immunologic, or behavioral disease, or infection or malignancy or concomitant illness or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risks for receiving the study drugs or a medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the participant's ability to comply with the protocol required testing or procedures or compromise the participant's wellbeing, safety, or clinical interpretability.
* Exposure to gene therapy, investigational medication, or other protocol-specified treatment within the protocol specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests.

Note: Other inclusion or exclusion criteria could apply.

Ages: 4 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression as Measured by Western Blot Adjusted by Muscle Content | Baseline, Week 12
Change From Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Expression in Biopsied Muscle as Measured by Immunofluorescence (IF) Fiber Intensity | Baseline, Week 12
Change From Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Expression in Biopsied Muscle as Measured by IF Percent Dystrophin-positive Fibers (PDPF) | Baseline, Week 12
Mean Concentration of Vector Genome Copies Using Polymerase Chain Reaction in Muscle Tissue Biopsy, After Delandistrogene Moxeparvovec Administration | Week 12

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Imlifidase | Up to Day 7
Total IgG in Serum After Imlifidase Administration | Up to Week 12
rAAVrh74 Antibody Titers After Imlifidase Administration | Up to Hour 120
Concentration of Vector Genome Copies Using Polymerase Chain Reaction in Serum, After Delandistrogene Moxeparvovec Administration | Up to Day 7
Number of Participants with a Treatment Emergent Adverse Event (TEAE), Adverse Event of Special Interest (AESI), and Serious Adverse Event (SAE) | Up to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain